Official Title: The Effects of Sedatives on Tobacco Use Disorder

NCT03813121 Date: 1/15/21

PI (researcher): Merideth Addicott, PhD

Institution: University of Arkansas for Medical Sciences Sponsor: University of Arkansas for Medical Sciences

# **University of Arkansas for Medical Sciences Informed Consent Form**

- We are asking you to be in a research study.
- You do not have to be in the study.
- If you say yes, you can quit the study at any time.
- Please take as much time as you need to make your choice.
- You can still get your medical care from UAMS even if you are not in the study.
- During the study, we will tell you if we learn any new information that might affect whether you wish to stay in the study.

#### Why am I being asked to be in this research study?

- We want to learn more about how to help people who smoke tobacco in the future. This study does not provide a treatment for smoking.
- This study will help us learn more about whether an infusion of medication (that is, a medication given through a small tube attached to a needle inserted into a vein) is safe and well tolerated, has any side effects, and will affect smokers' tobacco use.
- We are asking people like you who smoke tobacco to help us. Up to 20 people aged 21-55 years old will be part of this study.
- During the study, you will receive a study drug given through a tube inserted in your vein. You will not know the specific drug, but you will be given a list of possible drugs (see below), one of which you will get. All drugs on the list are approved by the FDA, but not as a treatment for tobacco smoking.

#### What if I don't understand something?

- This form may have words you don't understand. The research staff will read it with you, if you like.
- You may ask as many questions as you like before you decide whether you want to be in this study.
- You are free to ask questions at any time before, during, or after you are in the study.

# How long will this study take and where will it take place?

PI (researcher): Merideth Addicott, PhD

Institution: University of Arkansas for Medical Sciences Sponsor: University of Arkansas for Medical Sciences

- The study will last about 4 weeks in total and will include:
  - ✓ a screening session (about 3 hours)
  - √ 2 7-day smoking diaries (to write down the number of cigarettes smoked each day)
  - ✓ 2 study days (about 2.5 hours each)
  - √ 1 drug infusion day (about 3 hours)
  - √ 1 follow-up visit (about 0.5 hours)
  - ✓ You will also be asked to not smoke 2 times, for 10 hours each time.
- The study will take place at the Psychiatric Research Institute (PRI) at UAMS. The screening part, outpatient visits, and follow up interview will take place on the 4<sup>th</sup> floor of PRI. The drug infusion will take place on the 5<sup>th</sup> or 6<sup>th</sup> floor of PRI.

#### What if I say yes, I want to be in this study?

You will be screened to make sure you qualify to be in the study.

- The screening will include:
  - ✓ medical history
  - √ physical exam
  - ✓ mental health exam
  - ✓ routine blood tests
  - √ heart test (electrocardiogram)
  - ✓ breath tests for tobacco smoking and alcohol
  - ✓ urine (pee) tests (1 test will tell us what drugs you may have used)
  - ✓ women will also have a pregnancy test
  - We will not charge you for the screening.
  - You and your doctor can ask for screening results.
  - If you are healthy and smoke cigarettes every day, you can be in the study.

#### What will I have to do if I am in the study?

- You will be asked to take home a paper diary and record the number of cigarettes you smoke each day for 7 days. On the 7<sup>th</sup> day you will also answer questions about your mood over the past week.
- You will be asked to stop smoking for 10 hours overnight before coming to the first study day. This study day will occur in the morning and first you will answer questions about your mood. Then, you will be offered a small amount of money to not smoke

PI (researcher): Merideth Addicott, PhD

Institution: University of Arkansas for Medical Sciences Sponsor: University of Arkansas for Medical Sciences

up to an additional 50 minutes. Lastly you will be allowed to smoke and will answer more questions about your mood.

- On the second study day, you will be given study medication through a tube inserted in your arm (infusion). You will be asked to not eat or drink anything besides water for about 7 hours before the study day, and during the 3-hour study day. You will not be allowed to smoke during the study day.
- A doctor will first examine you to make sure you can safely have the procedure. Your blood pressure and your body's ability to take in oxygen from the air you breathe will be taken. If the doctor says the medication infusion can happen, a needle will be put in the vein in your arm and salt water will be put through the tube, followed by the medication over a 20-minute period. The medication will be one of these:

| Name of study medication | What the FDA has approved the medication to d |
|---|---|
| placebo | no active medication |
| ketamine | block pain, help you sleep, block memory |
| midazolam | help you sleep, decrease anxiety, block memory |

- You will be given only one medication on the list and no medication that is not on the list. We cannot tell you which drug you will receive now, because it may affect the way you answer questions during the study sessions. If you wish to know the actual drug tested, we can give you that information after all subjects have finished the study by mailing the name of the medication within 2 months after the study ends to the address we have on file for you.
- At least 1 out of 3 participants will receive placebo (no active medication) or one of the active drugs. This is decided randomly (by chance).
- After the infusion, the doctor or nurse will watch you for a couple of hours and will measure your vital signs (such as pulse and blood pressure) every 15 to 60 minutes. After 3 hours, you will be allowed to go home. Someone else must drive you home. If no one can drive you to and from the hospital, a taxi will be provided at no cost to you. You will be asked to stop smoking for 10 hours overnight before coming to the third study day, scheduled the following morning.

PI (researcher): Merideth Addicott, PhD

Institution: University of Arkansas for Medical Sciences Sponsor: University of Arkansas for Medical Sciences

The third study day is identical to the first study day, you will answer questions about your mood and you will be offered money to not smoke an additional 50 minutes. When this is completed, you may continue smoking as usual.

You will be given a second 7-day smoking diary on the third study day. About 8 days after the third study day, you will attend a follow-up visit. During the visit you will give a breath sample to test for smoking and answer questions about your symptoms and mood.

#### Who will see the information about me that is collected?

- The study team will know your name and have access to your information. Medical personnel will know your name, but cannot access research documents.
- We will do our best to make sure no one outside the study knows you are part of the study.
  - ✓ All research data will be labeled with a code that is linked to your name on a master list that is kept in a locked file cabinet in a secured room.
  - ✓ When we share the results of the study in presentation, posters and articles, we will not include your name or any other details that might identify you.
- This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means researchers cannot be made to release information or biospecimens, even by a court order or subpoena, unless you have given consent for this use. This is not a guarantee. Your information might be released if:
  - ✓ You have a disease others could catch from you (such as TB or HIV)
  - ✓ Researchers report current abuse (such as child or adult abuse) you may be involved in
  - ✓ Researchers think you are in danger of hurting yourself or others
  - ✓ A federal agency or UAMS office asks for information for the purposes of auditing or program evaluation

The Certificate of Confidentiality does not mean you cannot voluntarily release information about your involvement in this research.

- Researchers may also give medical information without your permission in the event of an emergency.
- There are also people who make sure the study is run the right way. These people may see information from the study about you. They are:
  - ✓ OHRP (Office for Human Research Protections), a federal agency
  - ✓ UAMS Institutional Review Board

PI (researcher): Merideth Addicott, PhD

Institution: University of Arkansas for Medical Sciences Sponsor: University of Arkansas for Medical Sciences

- ✓ Other UAMS institutional oversight offices
- ✓ FDA (Food and Drug Administration)
- State law does require that we tell the authorities if we learn
  - ✓ about possible child or adult abuse
  - ✓ that you might hurt yourself or someone else

## Where and how long will my information and samples be kept?

- We will code your information and study samples and keep the code in a locked file.
- Research records will be kept for up to 5 years after the study results are published.
- Only research staff members will have access to the code for your information.
- We will not put information about you from the study in your medical record.

#### What if I say no, I do not want to be in this study?

- Nothing bad will happen.
- You can still get medical care at UAMS.

#### What are alternatives to being in this study?

• If you do not wish to participate in this study, your alternative is not to participate.

#### What happens if I say yes, but change my mind later?

- Being in the study is completely up to you. You may leave the study at any time.
- If you decide to not be in the study (now or later), nothing bad will happen.
- You can still get health care at UAMS.
- If you decide to stop being in the study, call the research staff at 501-526-8462.
- If you change your mind after the study started, your lab samples and study records will stay in the study files.

#### Can I be taken out of the study even if I want to continue?

Yes, the study doctor (or head researcher) can take you out of the study if:

- You do not follow study instructions.
- It is not in your best interest to continue.

PI (researcher): Merideth Addicott, PhD

Institution: University of Arkansas for Medical Sciences Sponsor: University of Arkansas for Medical Sciences

- The study is stopped for any reason.
- You do not behave properly during the study visits.
- For any reason that may not be known at this time.

# If I stop being in the study, what will happen to any information or samples collected from me in the study?

We will not be able to take your information or samples out of the study after it has started.

# Will my information or samples from the study be used for anything else, including future research?

No. Your information and samples will be used only in this study. No study information will be collected about you after your participation has ended.

## Will it cost me anything to be in the study?

The study will not cost you anything.

#### Will I be paid?

Yes. We will give you money to thank you for your time as follows:

| Day(s) or Procedure | Amount per Day or Procedure |
|------------------------------------------------|-----------------------------|
| 7-day smoking diary | \$10 |
| Study days #1 and #3 (not the screening visit) | \$75 |
| Bonus for not smoking on study days | up to \$14 |
| Drug infusion | \$100 |
| Follow up Interview | \$10 |
| Completion bonus | \$100 |
| Total for all study visits/procedures | \$408 |

PI (researcher): Merideth Addicott, PhD

Institution: University of Arkansas for Medical Sciences Sponsor: University of Arkansas for Medical Sciences

You can earn up to \$408 for being in this study. You will be paid the full amount earned by check at the follow-up visit. If you do not come to all visits or drop out before the end of the study, you will get a check for the amount you had earned. If you do not come to the follow up visit, the check will be mailed to you at the address you give us.

If you receive more than \$600 in one year (January-December) from UAMS, UAMS may report the amount earned to the Internal Revenue Service (IRS) and send you a tax form, if required by law.

## Will being in this study help me in any way?

This study is not expected to help you, but what is learned from the study might help others who want treatment for their tobacco use.

## What are the risks of being in this study?

The main risks:

## Taking ketamine can cause

- ✓ changes in breathing rate
- ✓ problems seeing
- changes in heart rate and bloodpressure
- ✓ muscle jerks
- ✓ decreased hunger
- ✓ nausea
- √ vomiting
- ✓ uneasiness

- ✓ make tobacco withdrawal worse
- √ desire to use ketamine
- pleasant or unpleasant dreamlike states
- √ vivid imagery
- √ hallucinations
- ✓ confusion
- ✓ excitement
- ✓ irrational behavior

Ketamine may increase the strength of prescription painkillers for a short while.

## Taking midazolam can cause

- √ changes in breathing rate
- √ sleepiness
- √ difficulty remembering

- √ anxiousness
- √ nervous excitement
- ✓ changes in blood pressure and

Version 8 1/15/21 Page 7

PI (researcher): Merideth Addicott, PhD

Institution: University of Arkansas for Medical Sciences Sponsor: University of Arkansas for Medical Sciences

heart rate ✓ vomiting ✓ nausea ✓ headache

## Withdrawal from smoking can cause

| ✓ | anxiety | ✓ | increased | ✓ | insomnia |
|---|---------------|---|----------------|---|-----------------|
| ✓ | difficulty | | appetite | ✓ | irritability, |
| | concentrating | ✓ | restlessness | | frustration, or |
| | | ✓ | depressed mood | | anger |

These symptoms can be unpleasant, are not dangerous and only last for a while.

#### Other risks or inconveniences

- ✓ You may feel pain and get a bruise from the blood draw or the needle that is put in the vein of your arm. You may feel faint. When liquid is sent to your arm through the tube, you may feel pain.
- ✓ Someone could find out that you were in the study and learn something about you that you did not want others to know. We will do our best to protect your privacy.
- ✓ The questions could make you sad or upset.
- ✓ This study may involve risks that are not currently known.

## WOMEN PLEASE NOTE: This research may have bad effects on an unborn fetus.

- ✓ Do not be in the study if you are pregnant or breastfeeding.
- ✓ We must do a test to make sure you are not pregnant before letting you in the study.
- ✓ If you agree to be in the study, you agree to not get pregnant and to use birth control during the study.

# What if I get sick or hurt while I'm in this study?

- If you are hurt by being in the study, you may be treated. You or your insurance will be charged for this treatment. It may include
  - √ first aid
  - ✓ emergency treatment
  - √ follow-up care
- If you get hurt when you are here for the study we will help you get the care you need.

PI (researcher): Merideth Addicott, PhD

Institution: University of Arkansas for Medical Sciences Sponsor: University of Arkansas for Medical Sciences

- If you get hurt or sick during the study when you are not here, call your doctor or 911 in an emergency.
- If you think being sick has to do with being in the study
  - ✓ tell the ER staff or your doctor about the study
  - ✓ give the name of the study and copy of this form if you have it
  - ✓ call the study doctor, Dr. Lide, as soon as you can

#### What if new information comes up about the study?

- We will call you or send you a letter.
- We will tell you about anything that might change your mind about being in the study.

#### Where can I find more information about this clinical trial?

This is clinical trial number NCT03813121. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### Who do I call if I have questions about the study?

- Dr. Addicott at or one of the study doctors at
- UAMS Institutional Review Board (IRB) representative at
  - √ have questions about your rights as a study subject
  - √ have questions concerning a research-related injury
  - ✓ can't reach the study team
  - ✓ need to speak to someone not directly involved with this study

For more information go to

## What should I do if I want to be in the study?

Sign this form. We will give you a copy of the form to keep.

## By signing the document I am saying:

- I understand that joining this study is voluntary.
- I agree to be in the study.

PI (researcher): Merideth Addicott, PhD

Institution: University of Arkansas for Medical Sciences Sponsor: University of Arkansas for Medical Sciences

- Someone talked with me about the information in this document and answered all my questions.
- I have been asked if I wish to talk directly to the head researcher or study doctor.

#### I know that:

- I can stop answering questions at any time and nothing will happen to me.
- I can call the office that supervises research (UAMS IRB) at the study or about my rights.
- My decision will not change my medical care at UAMS.
- I do not give up any of my rights by signing this form.
- The purpose and voluntary nature of this study, as well as the potential benefits and risks that are involved have been explained to me. I have been able to ask questions and express concerns, which have been satisfactorily responded to by the study team. I understand that I have waived no rights by signing this consent form.
- I have been told that I will be given a signed copy of this consent form.

## I agree to be part of this study:

| Your name (please print) | Your signature |
|---|---|
| Date | |
| Name of person obtaining consent (please print) | Signature of person obtaining consent |
| <br>Date | |